CLINICAL TRIAL: NCT04238039
Title: Five Years Follow up: Add on Intravenous Ketamine for Major Depressive Disorder
Brief Title: Ketamine Long Therm Follow Up Study
Acronym: ket_Fol_Up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Revital Amiaz, Head of Psychiatry Department B, The Chaim Sheba Medical Center
Other Study IDs: 5826-18-SMC
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Followin Ketamine Treatment
Keywords: Major Depressive Disorder, ketamine, follow up, relapse
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Results of the study and of 5 years follow up of depressed patients who participated in the study during 2014-2015. We will locate the participants and will interview them will use the same questionnaires to evaluate their depressive symptoms. We will also measure the time to relapse.

DETAILED DESCRIPTION:
Anamnestic data will be collected from the patients, in addition, depressive symptoms will be measured using Montgomery Asberg Depression Scale (MADRAS). In addition, the Clinical Global Severity Scale (CGI-S) and Clinical Global Improvement (CGI-I) were performed 2 hours after treatment. In addition, we performed to prolong the time to relapse in this patient.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the ketamine study

Exclusion Criteria:

-

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the ketamine study
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to relapse | 5 years
  Medications

CONTACTS AND LOCATIONS:
Locations (1):
- Revital Amiaz, Ramat Gan, RI, Israel